CLINICAL TRIAL: NCT00305396
Title: Calcineurin Inhibitor Avoidance With Thymoglobulin and Sirolimus in Kidney Transplant Recipients.
Brief Title: Calcineurin Inhibitor Avoidance With Thymoglobulin and Sirolimus in Kidney Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 031041
Record Dates: First submitted 2006-03-20; First posted 2006-03-21 (Estimated); Last update posted 2006-03-21 (Estimated); Status verified 2006-03

CONDITIONS: Kidney Transplantation
Keywords: Kidney transplantation; immunosuppression; sirolimus; Thymoglobulin
MeSH Terms: interventions — Sirolimus

INTERVENTIONS:
Drug: Sirolimus

SUMMARY:
A prospective, single center, open-label, randomized trial of Thymoglobulin induction and sirolimus, prednisone, and mycophenolate mofetil versus Thymoglobulin induction and tacrolimus, prednisone, and mycophenolate mofetil in non-HLA identical living or deceased donor kidney transplant recipients.

DETAILED DESCRIPTION:
Calcineurin inhibitor-associated nephrotoxicity may exacerbate chronic allograft nephropathy and reduce long-term kidney graft survival. Complete avoidance of calcineurin inhibitors may improve graft function as measured by serum creatinine and calculated GFR and improve long-term outcomes following kidney transplantation. We conducted a prospective, randomized, single-center study comparing sirolimus versus tacrolimus in kidney transplantation. Primary cadaver of non-HLA identical living donor recipients are randomized to received either sirolimus 5 mg QD (target level 8-12 ng/ml) or tacrolimus 0.075 mg/kg BID (target level 8-12 ng/ml). All patients also received Thymoglobulin 1.5 mg/kg x 4 doses, mycophenolate 1 gm BID, and prednisone. Main outcome measures are patient and graft survival, biopsy-proven acute rejection, serum creatinine, hyperlipidemia, post-transplant diabetes, and surgical and wound complications.

ELIGIBILITY:
Inclusion Criteria:

Primary cadaver or non-HLA identical living donor kidney transplant. -

Exclusion Criteria:

HIV HCV Pregnancy Age < 18 years Malignancy

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2004-04; Study Completion 2005-03

PRIMARY OUTCOMES:
Patient and graft survival
Biopsy proven acute rejection
Serum creatinine

SECONDARY OUTCOMES:
Hyperlipidemia
post-transplant diabetes
wound infections
lymphoceles

CONTACTS AND LOCATIONS:
Overall Officials: A. Tarik Kizilisik, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center/Nashville VA, Nashville, Tennessee, United States

REFERENCES:
- [Background] Flechner SM, Goldfarb D, Modlin C, Feng J, Krishnamurthi V, Mastroianni B, Savas K, Cook DJ, Novick AC. Kidney transplantation without calcineurin inhibitor drugs: a prospective, randomized trial of sirolimus versus cyclosporine. Transplantation. 2002 Oct 27;74(8):1070-6. doi: 10.1097/00007890-200210270-00002. PMID 12438948